CLINICAL TRIAL: NCT05531292
Title: PROOF-OF-CONCEPT STUDY FOR NEW INTRAOCULAR LENS, MODEL C0002
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Surgical Vision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PCOL106APV2
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Cataracts
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Lens (Experimental): investigational IOL Model C0002
  Interventions: Device: Model C0002
- Control Lens (Active Comparator): control IOL Model ZCB00/DCB00
  Interventions: Device: Model ZCB00/DCB00

INTERVENTIONS:
Device: Model C0002 — Eligible subjects will be randomized in a 1:1 ratio to the investigational IOL Model C0002 in both eyes for the duration of the study.
  Arms: Study Lens
Device: Model ZCB00/DCB00 — Eligible subjects will be randomized in a 1:1 ratio to the control IOL Model ZCB00 in both eyes for the duration of the study.
  Arms: Control Lens

SUMMARY:
Prospective, two-arm, randomized, bilateral, subject/evaluator-masked clinical study to evaluate the distance visual acuity, peripheral refractive error and functional vision of the EPV IOL compared to a standard monofocal control IOL.

ELIGIBILITY:
Inclusion Criteria:

1. Age of study population between 60-75 years;
2. Bilateral cataracts for which cataract extraction and posterior chamber IOL implantation have been planned for both eyes;
3. Cataractous lens changes, as demonstrated by best-corrected distance visual acuity (BCDVA) of 0.50 decimal or worse (6/12 or 20/40 Snellen) either with or without a glare source present (e.g., Brightness Acuity Tester) or with significant cataract related visual symptoms in the opinion of the investigator;
4. Potential postoperative best-corrected distance visual acuity (BCDVA) of 0.66 decimal (6/9 or 20/30 Snellen) or better;
5. Drives a car at least 1-2 times per month;
6. Corneal astigmatism:

   1. Normal corneal topography
   2. Predicted postoperative residual refractive cylinder based on a toric IOL calculator, taking surgically induced astigmatism (SIA) into account and using the posterior corneal astigmatism (PCA) option, must be less than 1.00 D in both eyes.
7. Clear intraocular media other than cataract in each eye;
8. Availability, willingness, sufficient cognitive awareness to comply with examination procedures;
9. Signed informed consent and HIPAA authorization or equivalent documentation necessary to comply with applicable privacy laws pertaining to medical treatment in the governing countries;
10. Ability to understand, read, and write in French.

Exclusion Criteria:

1. Requiring an intraocular lens power needed to achieve emmetropia (spherical equivalent ± 0.50 D) outside the available range of +18.0 D to +30.0 D for the Model C0002 IOL or +16.5 D to +27.5 D for the Model ZCB00 IOL;
2. Pupil abnormalities (non-reactive, fixed pupils, or abnormally-shaped pupils);
3. Irregular corneal astigmatism;
4. Recent ocular trauma or ocular surgery that is not resolved/stable or may affect visual outcomes or increase risk to the subject;
5. Prior corneal refractive (LASIK, LASEK, RK, PRK, etc.) or intraocular surgery;
6. Subjects who may be expected to require retinal laser treatment during the study;
7. Corneal abnormalities such as stromal, epithelial or endothelial dystrophies that are predicted to cause visual acuity losses to a level of worse than 0.66 decimal (6/9 or 20/30 Snellen) during the study;
8. Inability to achieve keratometric corneal stability preoperatively as a result of recent contact lens usage;
9. Subjects with diagnosed degenerative visual disorders (e.g., retinal disorders such as macular degeneration) that are predicted to cause visual acuity losses to a level worse than 0.66 decimal (6/9 or 20/30 Snellen) during the study;
10. Subjects with conditions associated with increased risk of zonular rupture, including capsular or zonular abnormalities that may lead to IOL decentration or tilt, such as pseudoexfoliation, trauma, or posterior capsule defects;
11. Use of systemic or ocular medications that may affect vision;
12. Prior, current, or anticipated use during the course of the study of tamsulosin or silodosin (e.g., Flomax, Flomaxtra, Rapaflo) that may, in the opinion of the investigator, confound the outcomes or increase the risk to the subject (e.g., poor dilation or a lack of adequate iris structure to perform standard cataract surgery);
13. Inability to focus or fixate for prolonged periods of time (e.g., due to strabismus, nystagmus, etc.);
14. Poorly-controlled diabetes;
15. Acute, chronic, or uncontrolled systemic or ocular disease or illness that, in the opinion of the investigator, would increase the operative risk or confound the outcomes of the study (e.g., immunocompromised, connective tissue disease, suspected glaucoma, glaucomatous changes in the fundus or visual field, ocular inflammation, etc.); NOTE: Controlled ocular hypertension without glaucomatous changes (optic nerve cupping and visual field loss) is acceptable.
16. Neurological or neurodegenerative disorders that affect locomotion and cognitive function (e.g., Muscular disorders, Parkinson's disease, Alzheimer's disease etc.);
17. Use of mobility aids, any injury or condition that may affect walking;
18. Subject has condition(s) associated with the fluctuation of hormones that could lead to refractive changes;
19. Concurrent participation in any other clinical trial or participation within 30 days prior to the preoperative visit.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2022-11-22 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Postoperative Refractive Error | within 14 days of completion of 1-month follow-up
  Ocular refractive error, including defocus and astigmatism, will be measured using an autorefractor instrument.
MONOCULAR, PHOTOPIC BCDVA AT 4 M | within 14 days of completion of 1-month follow-up
  Distance visual acuity will be measured postoperatively at 100% contrast under photopic lighting conditions (85 cd/m2, 80-110 cd/m2 acceptable).

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Surgical Vision, Inc. Clinical Trial, Study Director — Johnson & Johnson Surgical Vision, Inc.
Locations (2):
- France (2):
  - Centre Hospitalier National d'Ophtalmologie, Paris, Île-de-France Region
  - Rothschild Foundation Hospital, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu